CLINICAL TRIAL: NCT06217562
Title: Vasopressin for Septic Shock Pragmatic Trial
Acronym: VASSPR
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Intermountain Health Care, Inc. (Other)
Collaborators: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 1052518
Record Dates: First submitted 2024-01-09; First posted 2024-01-22 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Septic Shock
Keywords: Vasopressin; Vasopressors; Treatment strategy
MeSH Terms: conditions — Shock, Septic; Diabetes Insipidus | interventions — Vasopressins

STUDY DESIGN:
Intervention Model Description: Pragmatic embedded cluster-randomized cluster-crossover comparative effectiveness trial. Study hospitals will be assigned to a vasopressin-initiation strategy (cluster randomized) and the hospital will then alternate monthly between the tested vasopressin-initiation strategies in a randomized sequence (cluster-crossover).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Septic shock treatment strategy involving a lower threshold for vasopressin initiation (Active Comparator): Recommended strategy for treatment of septic shock includes initiation of fixed-dose IV vasopressin (1.8 units/hour) as a second-line vasopressor if the combined norepinephrine-equivalent dose of other vasopressors reaches ≥0.1 micrograms/kilogram/minute (mcg/kg/min). Use of the recommended treatment strategy (via entry of an order for threshold-based vasopressin initiation) or an alternative treatment strategy is at the discretion of patients' treating clinical team.
  Interventions: Drug: Vasopressin; Other: Recommendation to use a lower initiation threshold for vasopressin
- Septic shock treatment strategy involving a higher threshold for vasopressin initiation (Active Comparator): Recommended strategy for treatment of septic shock includes initiation of fixed-dose IV vasopressin (1.8 units/hour) as a second-line vasopressor if the combined norepinephrine-equivalent dose of other vasopressors reaches ≥0.4 mcg/kg/min. Use of the recommended treatment strategy (via entry of an order for threshold-based vasopressin initiation) or an alternative treatment strategy is at the discretion of patients' treating clinical team.
  Interventions: Drug: Vasopressin; Other: Recommendation to use a higher initiation threshold for vasopressin

INTERVENTIONS:
Drug: Vasopressin — Intravenous vasopressin infusion added to first-line vasopressors. Recommended vasopressin dose is 1.8 units/hour (equivalent to 0.03 units/minute) at a fixed rate.
Other: Recommendation to use a lower initiation threshold for vasopressin — Recommended to initiate intravenous vasopressin infusion if the combined dose of other vasopressors reaches ≥0.1 mcg/kg/min of norepinephrine (or equivalent)
  Arms: Septic shock treatment strategy involving a lower threshold for vasopressin initiation
Other: Recommendation to use a higher initiation threshold for vasopressin — Recommended to initiate intravenous vasopressin infusion if the combined dose of other vasopressors reaches ≥0.4 mcg/kg/min of norepinephrine (or equivalent)
  Arms: Septic shock treatment strategy involving a higher threshold for vasopressin initiation

SUMMARY:
Life-threatening low blood pressure due to a serious infection is called "septic shock." Septic shock is treated with vasopressors, medications that raise blood pressure. Sometimes first-line vasopressors are inadequate, prompting addition of a second-line vasopressor called vasopressin. However, the threshold at which to start vasopressin remains unclear. This pragmatic, cluster-randomized, cluster-crossover trial will evaluate two different strategies for septic shock treatment commonly used in current practice, comparing a lower versus a higher threshold for adding vasopressin to first-line vasopressors.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Admitted to a study hospital emergency department (ED) or inpatient care unit
3. Administration of vasopressor(s) for septic shock

Exclusion Criteria: None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2050 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
28-day all-cause mortality | 28 days
  Death on or before study day 28

SECONDARY OUTCOMES:
Renal replacement therapy-free days to day 28 | 28 days
  Number of days between day 28 and the end of the last period of renal replacement therapy prior to day 28. Death on or before day 28 will be assigned a value of -1. For patients with baseline end-stage renal failure on dialysis prior to the index hospitalization, potential values for this ordinal outcome will be 0 or -1.

OTHER OUTCOMES:
In-hospital all-cause mortality | From onset of septic shock to hospital discharge, an average of 10 days
  Death prior to discharge from the hospital
90-day all-cause mortality | 90 days
  Death on or before study day 90
Vasopressor-free days to day 28 | 28 days
  Number of days between day 28 and the end of the last period of vasopressor therapy prior to day 28. Death on or before day 28 will be assigned a value of -1.
Incidence of new renal replacement therapy | From onset of septic shock until hospital discharge, an average of 10 days
  New receipt of renal replacement therapy after onset of septic shock. Patients receiving renal replacement therapy prior to enrollment are excluded from this outcome.
Intensive care unit-free days to day 28 | 28 days
  Number of days between day 28 and the end of the last period of intensive care unit admission prior to day 28. Death on or before day 28 will be assigned a value of -1.
Hospital-free days to day 28 | 28 days
  Number of days between day 28 and the end of the last period of hospital admission prior to day 28. Death on or before day 28 will be assigned a value of -1.
Incidence of acute coronary syndrome | From onset of septic shock until hospital discharge, an average of 10 days
  Documented new-onset clinical diagnosis of acute coronary syndrome or myocardial infarction
Incidence of mesenteric ischemia | From onset of septic shock until hospital discharge, an average of 10 days
  Documented new-onset clinical diagnosis of mesenteric ischemia
Incidence of soft tissue ischemia | From onset of septic shock until hospital discharge, an average of 10 days
  Documented new-onset clinical diagnosis of extremity, nose, or ear ischemia
Incidence of vasopressor extravasation | From onset of septic shock until hospital discharge, an average of 10 days
  Documented clinical diagnosis of vasopressor extravasation
Incidence of clinically-significant arrhythmia | From onset of septic shock until hospital discharge, an average of 10 days
  Documented clinical diagnosis of clinically-significant arrhythmia (sustained ventricular tachycardia, reentrant [supraventricular] tachycardia, atrial arrhythmia with rapid ventricular response requiring intervention, or new-onset atrial fibrillation or flutter)
Incidence of cardiogenic shock | From onset of septic shock until hospital discharge, an average of 10 days
  Documented clinical diagnosis of cardiogenic shock
Incidence of cardiac arrest | From onset of septic shock until hospital discharge, an average of 10 days
  Documented occurrence of a cardiac arrest with administration of chest compressions or defibrillation
Incidence of severe hyponatremia | From onset of septic shock until hospital discharge, an average of 10 days
  New-onset severe hyponatremia (serum sodium <120 milliequivalents/liter)
Maximum lactate | 7 days
  Maximum lactate value (millimoles/liter) from enrollment through study day 7
Incidence of abnormal troponin | 7 days
  Serum troponin above the upper limit of normal for assay in interval from enrollment through study day 7

CONTACTS AND LOCATIONS:
Overall Officials: Ithan Peltan, MD, MSc, Principal Investigator — Intermountain Health
Locations (13):
- United States (13):
  - Cassia Regional Hospital, Burley, Idaho
  - American Fork Hospital, American Fork, Utah
  - Cedar City Hospital, Cedar City, Utah
  - Layton Hospital, Layton, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital, Ogden, Utah
  - Park City Hospital, Park City, Utah
  - Utah Valley Hospital, Provo, Utah
  - Riverton Hospital, Riverton, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Alta View Hospital, Sandy City, Utah
  - St. George Regional Hospital, St. George, Utah

IPD SHARING:
Plan to Share IPD: Yes
In order to protect patient privacy and comply with relevant regulations, identified data will be unavailable. Requests for deidentified data from qualified researchers with appropriate ethics board approvals and relevant data use agreements will be processed by the Intermountain Office of Research, officeofresearch@imail.org.
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Derived] Peltan ID, Groat D, Jacobs JR, Tillman EH, Brintz BJ, Chauv S, Beesley SJ, Edwards JH, Arizmendez N, Hirshberg EL, Carr JR, Lanspa MJ, Bledsoe JR, Smith AT, Schneider H, Hu P, Moores Todd TD, Klippel C, Semler MW, Casey JW, Grissom CK, Brown SM, Leither LM. Protocol and Statistical Analysis Plan for the Vasopressin for Septic Shock Pragmatic (VASSPR) Cluster-Crossover Randomized Trial. CHEST Crit Care. 2025 Dec;3(4):100178. doi: 10.1016/j.chstcc.2025.100178. Epub 2025 Nov 12. PMID 41552411